CLINICAL TRIAL: NCT01486043
Title: Metformin as an Adjunctive Therapy For Transient Hyperglycemia in Patients With Acute Lymphoblastic Leukemia During Induction Chemotherapy
Brief Title: Metformin and Transient Hyperglycemia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The research project was terminated due to lower than projected patient recruitment within the period of time allowed for the study.
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Dr. Jamie R. Wood, Assistant Professor of Clinical Pediatrics; Director of Clinical Diabetes Programs at Children's Hospital Los Angeles, University of Southern California, Keck School of Medicine, Children's Hospital Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCI-11-00295
Record Dates: First submitted 2011-11-30; First posted 2011-12-06 (Estimated); Results first posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Acute Lymphoblastic Leukemia; Hyperglycemia; Insulin Resistance; Diabetes Mellitus
Keywords: Induction chemotherapy; Transient hyperglycemia; Metformin; Acute lymphoblastic leukemia; Insulin resistance; Hyperglycemia; Insulin
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Hyperglycemia; Insulin Resistance; Diabetes Mellitus | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin and insulin therapy (Experimental): Up to 30-40 patients will be in the prospectively recruited treatment group, which will receive both metformin and insulin therapy for transient hyperglycemia
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — All subjects will be started on metformin 500 mg orally twice daily. The dose will be increased by 500 mg weekly as tolerated until subjects' blood glucoses are well controlled or until the patient reaches metformin 1000 mg PO BID.
  Other Names: Glucophage, Metformin HCl

SUMMARY:
The purpose of this study is to determine whether metformin is an effective adjunctive treatment for transient hyperglycemia in patients with acute lymphoblastic leukemia (ALL) undergoing induction chemotherapy

DETAILED DESCRIPTION:
ALL is the most common childhood cancer, representing one fourth of all cancers diagnosed under the age of 15 years. One of the most common side effects of ALL chemotherapy is transient hyperglycemia. Patients that develop this complication require treatment with insulin via injections to prevent severe medical complications such as dehydration, weight loss, ketoacidosis and life-threatening infections. Although insulin therapy is effective, it adds a lot of physical and psychological burden to patients because multiple daily insulin injections are required to achieve adequate blood glucose control.

In this pilot study, investigators aim to examine the effectiveness of metformin as an adjunctive treatment for transient hyperglycemia. Investigators will be comparing two groups of subjects (up to 40 subjects per group). Patients in the treatment group will be prospectively recruited, and they will be treated with metformin in addition to insulin therapy. Investigators will compare the treatment group to a historical control group acquired via chart review. These patients will have been treated with insulin alone.

Statistical comparison will be made between the two groups in terms of the length of insulin treatment, the total daily dose of insulin required, number of insulin injections, hemoglobin A1c level (measure of glycemic control over preceding 8- 12 weeks), and fructosamine level (measure of glycemic control over preceding 2-3 weeks).

Investigators hypothesize that the use of metformin will result in fewer numbers of insulin injections and fewer days of insulin therapy.

ELIGIBILITY:
Inclusion Criteria:

* ALL patients on induction chemotherapy who develop transient hyperglycemia(definition of transient hyperglycemia: random blood glucose > 200 mg/dL x 2)
* Adequate renal function (serum Cr < 1.5 mg/dL in males, < 1.2 mg/dL in females)
* Adequate hepatic function (AST < 5x upper limit of normal)

Exclusion Criteria:

* Patients with known diagnosis of diabetes or those that are already on oral hypoglycemic agents or insulin
* Allergy to metformin or any component of the formulation
* Patients with pancreatitis (lipase level > 300 Units/L)
* Patients with active infection (positive blood culture within 48 hours of study registration)
* Patients with hemodynamic instability (PICU status, need for vasopressors within 48 hours of study entry)
* Elevated hemoglobin A1c (greater than 6.0%)

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2011-12; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie R Wood, M.D., Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Background] Pui CH, Burghen GA, Bowman WP, Aur RJ. Risk factors for hyperglycemia in children with leukemia receiving L-asparaginase and prednisone. J Pediatr. 1981 Jul;99(1):46-50. doi: 10.1016/s0022-3476(81)80955-9. PMID 6454771
- [Background] Baillargeon J, Langevin AM, Mullins J, Ferry RJ Jr, DeAngulo G, Thomas PJ, Estrada J, Pitney A, Pollock BH. Transient hyperglycemia in Hispanic children with acute lymphoblastic leukemia. Pediatr Blood Cancer. 2005 Dec;45(7):960-3. doi: 10.1002/pbc.20320. PMID 15700246
- [Background] Lowas SR, Marks D, Malempati S. Prevalence of transient hyperglycemia during induction chemotherapy for pediatric acute lymphoblastic leukemia. Pediatr Blood Cancer. 2009 Jul;52(7):814-8. doi: 10.1002/pbc.21980. PMID 19260096
- [Background] Howard SC, Pui CH. Endocrine complications in pediatric patients with acute lymphoblastic leukemia. Blood Rev. 2002 Dec;16(4):225-43. doi: 10.1016/s0268-960x(02)00042-5. PMID 12350366
- [Background] Sonabend RY, McKay SV, Okcu MF, Yan J, Haymond MW, Margolin JF. Hyperglycemia during induction therapy is associated with poorer survival in children with acute lymphocytic leukemia. J Pediatr. 2009 Jul;155(1):73-8. doi: 10.1016/j.jpeds.2009.01.072. Epub 2009 Apr 25. PMID 19394046

RESULTS

PARTICIPANT FLOW:
Groups:
- Metformin and Insulin Therapy: For the prospectively recruited arm (metformin plus insulin therapy), a total of 4 subjects were recruited. Two subjects were withdrawn from the study after laboratory studies revealed liver enzymes (AST) levels that were above that allowed for the study at the time. An additional 2 subjects were recruited in the study.
  For the retrospective chart review portion of our study, 12 patients were included after conducting chart review of cases from January 2007 to August 2011.
Period: Overall Study
Arm/Group | Metformin and Insulin Therapy
Started | 4
Completed | 2 (Study terminated due to insufficient recruitment)
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Metformin and Insulin Therapy: Patients receiving metformin and insulin therapy.
Arm/Group | Metformin and Insulin Therapy
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 13.5 [12 to 15]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 2
Hemoglobin A1C [Mean (Full Range); unit: %] | 5.8 [5.5 to 6]
Fructosamine [Mean (Full Range); unit: uM] | 193 [178 to 207]
# of Day of Induction at Onset of Hyperglycemia [Mean (Full Range); unit: days] | 2 [2 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Length of Insulin Therapy (Days)
Time Frame: During the 30 days of induction chemotherapy (plus or minus 2 weeks)
Measure: Mean (Full Range); unit: days
Arm/Group | Metformin and Insulin Therapy
Number analyzed (Participants) | 2
days | 7.5 [0 to 15]

2. Secondary Outcome: Serum Fructosamine Level
Time Frame: At 1 month
Measure: Mean (Full Range); unit: uM
Arm/Group | Metformin and Insulin Therapy
Number analyzed (Participants) | 2
uM | 190 [182 to 198]

3. Secondary Outcome: Hemoglobin A1c
Time Frame: At 1 month
Measure: Mean (Full Range); unit: percent of hemoglobin
Arm/Group | Metformin and Insulin Therapy
Number analyzed (Participants) | 2
percent of hemoglobin | 4.8 [4.3 to 5.3]

ADVERSE EVENTS:
Arm/Group | Metformin and Insulin Therapy
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No